CLINICAL TRIAL: NCT02872545
Title: Influence of Patient Position on Attenuation Artifacts Observed in D-SPECT Camera Myocardial Tomoscintigraphy
Acronym: D-SPECT BIKER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A00378-43
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Attenuation Artifact; Myocardial Tomoscintigraphy; Patient Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- forward tilted (Experimental): Patients with abnormal results at stress myocardial perfusion tomoscintigraphy will undergo a rest tomoscintigraphy. Acquisition will be done in forward tilted position
  Interventions: Procedure: Rest tomoscintigraphy in forward tilted; Procedure: Rest tomoscintigraphy in semi sitting position; Procedure: Rest tomoscintigraphy in dorsal decubitus position
- semi sitting (Other): Patients with abnormal results at stress myocardial perfusion tomoscintigraphy will undergo a rest tomoscintigraphy. Acquisition will be done in semi sitting
  Interventions: Procedure: Rest tomoscintigraphy in forward tilted; Procedure: Rest tomoscintigraphy in semi sitting position
- dorsal decubitus (Other): Patients with abnormal results at stress myocardial perfusion tomoscintigraphy will undergo a rest tomoscintigraphy. Acquisition will be done in dorsal decubitus
  Interventions: Procedure: Rest tomoscintigraphy in forward tilted; Procedure: Rest tomoscintigraphy in dorsal decubitus position

INTERVENTIONS:
Procedure: Rest tomoscintigraphy in forward tilted — Rest tomoscintigraphy in forward tilted position
Procedure: Rest tomoscintigraphy in semi sitting position — Rest tomoscintigraphy in forward tilted position, followed by a second rest tomoscintigraphy in semi sitting position, after max 30 min
  Arms: forward tilted; semi sitting
Procedure: Rest tomoscintigraphy in dorsal decubitus position — Rest tomoscintigraphy in forward tilted position, followed by a second rest tomoscintigraphy in semi sitting position, after max 30 min
  Arms: dorsal decubitus; forward tilted

SUMMARY:
The purpose is to compare percentages of myocardial segments showing attenuation in patients in forward tilted position (biker position) or 2 conventional positions (dorsal decubitus or semi sitting) at acquisition with D-SPECT camera in myocardial tomoscintigraphy.

The hypothesis is that the percentage of myocardial segments with attenuation is significantly lower when acquisitions are made in forward tilted position (biker position).

The secondary purpose is to restrict this analysis to 3 cardiac regions most subject to attenuation artifacts (anterior, apical and inferobasal regions).

DETAILED DESCRIPTION:
Myocardial perfusion tomoscintigraphy is a very used technique for diagnosis and characterization of abnormalities of stress and rest myocardial perfusion (ischemia, infarction).

A common problem is attenuation artifacts that are due to tissue interposition attenuating radiation from some cardiac regions. These artifacts originate activity decreasing and thus perfusion abnormalities potentially in all walls of left ventricle, especially the inferior wall in men (attenuation by sub-diaphragmatic organs) and the anterior wall in women (attenuation by mammary glands). These artifacts are observed in rest and stress acquisitions and can lead to a wrong diagnosis of infarction.

Attenuation artifacts can be identified with analysis of contraction kinetics with "gated-SPECT" (normal kinetics and thus discordant with aspect of infarction). With D-SPECT camera some artifacts can be prevented with a 30-35° forward tilted position of acquisition. This position, also called biker position, can take cardiac area away from sub-diaphragmatic structures. It can also reduce the distance between heart and detection surface of camera and limit respiratory movements of thoracic wall.

In this study, patients with abnormal results at stress myocardial perfusion tomoscintigraphy will undergo a rest tomoscintigraphy. Acquisition will be done in forward tilted position and in one of 2 other positions: dorsal decubitus or semi sitting.

ELIGIBILITY:
Inclusion Criteria:

* Affiliation to social security
* Signed informed consent
* Previous clinical examination authorizing patient to undergo tomoscintigraphy
* Patient with abnormal results of stress tomoscintigraphy and needing a rest tomoscintigraphy
* Patient with sinus and regular cardiac rhythm
* Patient with stable clinical status (without signs of unstable cardiac or coronary failure, without uncontrolled hypertension under treatment)

Exclusion Criteria:

* Women of childbearing potential without effective contraception
* Evolutive pregnancy
* Breastfeeding patient
* Contraindication to tomoscintigraphy
* Patient with history of hypersensibility to tomography radiotracer STAMICIS® or one of components
* Patient in life-and-death emergency
* Patient with history of disorders possibly interfering with contractility
* Patient with normal results of stress tomoscintigraphy
* Person under legal protection or incapable to consent
* Person deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of myocardial segments classified with attenuation artifact | day 0
  With infarction aspect but normal contraction kinetics in Gated-SPECT analysis.
  Left ventricle is divided in 17 segments according to American Heart Association.

SECONDARY OUTCOMES:
Percentage of myocardial segments classified with attenuation artifact in anterior region | day 0
Percentage of myocardial segments classified with attenuation artifact in apical region | day 0
Percentage of myocardial segments classified with attenuation artifact in inferobasal region | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu PERRIN, Dr, Principal Investigator — Service de Médecine Nucléaire - CHRU de Nancy-Brabois - Vandoeuvre Lès Nancy
Locations (1):
- Service de Médecine Nucléaire - CHRU de Nancy-Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No